CLINICAL TRIAL: NCT07032077
Title: Phase II Clinical Trial on the Safety, Tolerability, and Efficacy of HRS-7058 Combined Anti-tumor Drugs in Subjects With Solid Tumors.
Brief Title: A Phase II Clinical Trial on the Safety, Tolerability, and Efficacy of HRS-7058 Combined Anti-tumor Drugs in Subjects With Solid Tumors.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-7058-201-CRC
Record Dates: First submitted 2025-06-13; First posted 2025-06-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-7058 (Experimental): HRS-7058 combimed with antitumor drugs
  Interventions: Drug: HRS-7058

INTERVENTIONS:
Drug: HRS-7058 — HRS-7058 combimed with antitumor drugs

SUMMARY:
This study aims to evaluate the safety and tolerability of HRS-7058 combined with antitumor drugs in subjects with solid tumors, and to determine the recommended dosage for Phase II. Evaluate the objective response rate of HRS-7058 in combination with anti-tumor drugs in subjects with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are capable of giving informed consent, have signed the informed consent form approved by the IRB/EC and noted the date, and are willing and able to comply with the treatment plan, visits, various examinations, and other procedural requirements.
2. Age must be between 18 and 75 years old (inclusive) when signing the informed consent form, gender is unrestricted.
3. ECOG score of 0 or 1;
4. Expected survival period ≥ 12 weeks;
5. Provide 5-15 pieces of tumor tissue blocks fixed in formalin and embedded in paraffin, or unstained tumor specimen slices. The samples should be archived within the first 3 years before treatment or freshly obtained (freshly obtained is preferred). Slices do not need to be provided during the dose escalation phase.
6. According to the RECIST v1.1 standard, there must be at least one measurable lesion.
7. The functions of important organs meet the standards (no blood components or cell growth factors were used for corrective treatment within 14 days prior to the first administration of the drug), and the examination results must be completed within 7 days before the first study treatment:
8. Female subjects of childbearing potential must undergo a serum pregnancy test within 7 days prior to the first dose, and the result must be negative (if the serum HCG test is positive, pregnancy causes must be ruled out and further discussion with the sponsor is required); and must not be breastfeeding. Female subjects of childbearing potential and male partners of female subjects of childbearing potential must agree to follow contraceptive requirements from the time of signing the informed consent until 5 months after the last administration of the study drug (for male subjects) or 8 months (for female subjects) (see "Methods of Contraception" in the study protocol attachments for details).

Exclusion Criteria:

1. Subjects with untreated or active CNS metastases, a history of meningeal metastasis, or current meningeal metastasis are not eligible for enrollment.
2. Start the study if the patient has received systemic anti-tumor treatment within 28 days prior to enrollment. If the patient has previously received small molecule targeted therapy, there must be an interval of at least 5 half-lives of that drug or 14 days, whichever is shorter, between the end of treatment and the first study treatment. If the patient has previously received traditional Chinese medicine or Chinese patent medicine for anti-tumor treatment, they may be enrolled if there is an interval of at least 14 days between the end of treatment and the first study treatment.
3. Palliative radiotherapy completed within 14 days before the first administration;
4. Unable to recover from the toxicity and/or complications of prior interventions to CTCAE ≤ Grade 1 (excluding conditions such as alopecia, Grade 2 peripheral neuropathy, and other situations deemed by the investigator not to affect the treatment with the investigational drug that meet the numerical requirements in the enrollment criteria);
5. Used strong CYP3A4 inhibitors and P-gp, BCRP inhibitors within 7 days prior to the first administration, or used strong CYP3A4 inducers within 14 days prior to the first administration;
6. Subjects with known or suspected interstitial pneumonia; those with significant pulmonary diseases impacting respiratory function in the three months prior to the first administration, including but not limited to idiopathic pulmonary fibrosis, organizing pneumonia/obliterative bronchiolitis, pulmonary embolism, severe asthma, severe COPD, moderate to severe obstructive/restrictive ventilatory dysfunction, or those with a history of undergoing total lung resection. Subjects who previously had grade 3 or higher interstitial pneumonia during treatment with immune checkpoint inhibitors are not allowed to enroll in this study.
7. Patients with serious cardiovascular and cerebrovascular diseases；
8. Patients with a history of or concurrent other malignant tumors, unless they have achieved complete remission for at least 5 years prior to screening and do not require other treatment for basal cell carcinoma or squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ, local prostate cancer after radical surgery, or ductal carcinoma in situ after radical surgery during the study period (hormonal treatment for non-metastatic prostate cancer or breast cancer is allowed);
9. Subjects who experienced severe infections within 28 days prior to the first dose of medication, including but not limited to infections requiring hospitalization, bacteremia, severe pneumonia, etc.; active infections treated with therapeutic intravenous antibiotics within 2 weeks prior to the start of study treatment;
10. Those with active pulmonary tuberculosis infection within 1 year before enrollment, or those with a history of active pulmonary tuberculosis infection over 1 year ago but have not received formal treatment.
11. Presence of active hepatitis B (HBV DNA above the normal upper limit of the research center) or hepatitis C (anti-HCV positive and HCV RNA above the lower limit of the analysis method); presence of active syphilis infection;
12. Live attenuated vaccine used within 28 days prior to the first administration of the study drug, or expected to use live attenuated vaccine during the anticipated treatment period;
13. Patients with a history of immune deficiency diseases, including positive HIV tests, other acquired or congenital immune deficiency diseases, and those with a history of allogeneic hematopoietic stem cell transplantation or organ transplantation;
14. Patients with third space fluid accumulation that cannot be controlled clinically, deemed unsuitable for enrollment by the investigator.
15. Patients with refractory nausea and vomiting, chronic gastrointestinal diseases, etc., leading to an inability to swallow HRS-7058, or with intestinal obstruction, undergoing intestinal resection, etc., leading to insufficient absorption of HRS-7058;
16. Patients who had significant clinically meaningful bleeding symptoms within 3 months before the first study medication, and those who had noticeable hemoptysis within 1 month before the first study medication with each episode of hemoptysis being ≥ 2.5ml;
17. Patients who have undergone other major surgeries excluding diagnosis or biopsy within 28 days prior to the first administration; those who have experienced traumatic minor surgeries (biopsy, endoscopy, and drainage) within 7 days prior to the first administration; patients with non-healing wounds (severe, non-healing or ruptured) or untreated fractures;
18. Women who are pregnant or breastfeeding (even if the subject's blood pregnancy test is negative, if the researcher considers the subject's other circumstances and believes there may be a possibility of pregnancy, they need to be excluded; breastfeeding women are also not allowed to stop breastfeeding in order to participate in this study);
19. Patients known to be allergic to any component of HRS-7058; patients with a known history of severe allergic reactions to the combined therapeutic antitumor drugs;
20. Patients with uncontrollable mental illnesses as well as known situations of alcoholism, drug abuse or misuse, and criminal detention that affect the completion of the research procedures.
21. According to the investigators' judgment, patients who may have other conditions that could increase the risk of participating in the study, interfere with the research results, or make them unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
The incidence of dose-limiting toxicities (DLT), the incidence and severity of adverse events (AE) (according to NCI-CTCAE v5.0 standards); | About 28 days
RP2D of HRS-7058 in combination with antitumor drugs in subjects with solid tumors. | From the first dose to the last visit, about 12 months

SECONDARY OUTCOMES:
The duration of response (DoR) evaluated by researchers in participants with solid tumors using HRS-7058 in combination with antitumodr | From the first dose to the last visit, about 12 months
The objective response rate (ORR) evaluated by researchers in participants with solid tumors using HRS-7058 in combination with antitumodr | From the first dose to the last visit, about 12 months
The disease control rate (DCR) evaluated by researchers in participants with solid tumors using HRS-7058 in combination with antitumodr | From the first dose to the last visit, about 12 months
The progression-free survival (PFS) evaluated by researchers in participants with solid tumors using HRS-7058 in combination with antitumodr | From the first dose to the last visit, about 12 months
The overall survival (OS) evaluated by researchers in participants with solid tumors using HRS-7058 in combination with antitumodr | From the first dose to the last visit, about 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided